CLINICAL TRIAL: NCT00425945
Title: Cardiovascular Effects of Pine Bark Extract
Brief Title: Understanding Pine Bark Extract as an Alternative Treatment (UPBEAT) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Funded by Toyo Shinyaku Co Ltd (Unknown)
Responsible Party: Principal Investigator, Randall Stafford, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 37698
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — pycnogenols; flavangenol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo delivered as four tablets matching the active product once daily orally.
  Interventions: Drug: Pine Bark Extract (Flavangenol®)
- Pine Bark Extract (Active Comparator): Flavangenol 200 mg Flavangenol is a brand of Pine Bark Extract manufactured by Toyo Shinyaku of Saga, Japan. Dosage delivered as four tablets, each containing 50 mg Flavangenol, all 4 tablets taken once per day.
  Interventions: Drug: Pine Bark Extract (Flavangenol®)

INTERVENTIONS:
Drug: Pine Bark Extract (Flavangenol®) — Flavangenol 200 mg per day. Flavangenol is a brand of pine bark extract manufactured by Toyo Shinyaku of Saga, Japan.
  Dosage delivered as four tablets, each containing 50 mg Flavangenol, all 4 tablets taken once per day orally for 12 weeks.
  Other Names: Pycnogenol (differing formulation)

SUMMARY:
The purpose of this study is to investigate the efficacy of Flavangenol® (Toyo Shinyaku, Japan), a pine bark extract, in lowering blood pressure and improving glycemic control and plasma lipoprotein profile.

DETAILED DESCRIPTION:
Cardiovascular disease is the number one cause of death in the Unites States. Our study tests the efficacy of pine bark extract in improving a number of cardiovascular disease risk factors. We are conducting a randomized, placebo-controlled, double-blind, parallel trial that will investigate the efficacy and safety of Flavangenol® (Toyo Shinyaku, Japan), a pine bark extract, among 130 study participants. These participants will be individuals at mildly or moderately elevated risk of cardiovascular disease (CVD) because of having prehypertension, excess body weight, and insulin insensitivity. We aim to determine (in order of priority):

1. The efficacy of Flavangenol in lowering blood pressure.
2. The efficacy of Flavangenol in improving glycemic control and plasma lipoprotein profile.
3. Changes in body weight, antioxidative capacity, anti-inflammatory markers, blood coagulation factors, and liver function tests in response to Flavangenol.
4. The safety of Flavangenol, as confirmation of past studies.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure between 125 and 159 mmHg and diastolic blood pressure (DBP) < 100 mmHg
* Body mass index (BMI) 25.0-34.9
* Triglycerides (TG) < 450 mg/dL
* Low Density Lipoprotein (LDL) < 200 mg/dL
* Fasting blood glucose (FBG) < 126 mg/dL

Exclusion Criteria:

* DBP > 95 mmHg
* LDL > 170 mg/dL
* TG > 300 mg/dL
* FBG > 110 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall S. Stafford MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Drieling RL, Gardner CD, Ma J, Ahn DK, Stafford RS. No beneficial effects of pine bark extract on cardiovascular disease risk factors. Arch Intern Med. 2010 Sep 27;170(17):1541-7. doi: 10.1001/archinternmed.2010.310. PMID 20876405

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the local community through the use of radio and print advertisements between January 31, 2007 and May 31, 2008.
Pre-assignment Details: Prior to randomization, participants were scheduled to complete two baseline visits three to seven days apart at the Stanford GCRC. Only those who successfully completed both baseline visits were randomized into the study.
Groups:
- Pine Bark Extract: 200 mg Flavangenol delivered once per day orally. Flavangenol is a brand of Pine Bark Extract manufactured by Toyo Shinyaku of Saga, Japan. Dosage delivered as four tablets 50 mg each; 4 tablets taken in the morning daily.
  Pine Bark Extract (Flavangenol®) : Flavangenol 200 mg per day. Flavangenol is a brand of pine bark extract manufactured by Toyo Shinyaku of Saga, Japan.
  Dosage delivered as four tablets, 50 mg per tablet, taken once per day orally for 12 weeks.
- Placebo: Placebo delivered as four tablets matching the active product; four tablets taken daily orally.
Period: Overall Study
Arm/Group | Pine Bark Extract | Placebo
Started | 64 | 66
Completed | 60 | 61
Not Completed | 4 | 5
Not completed — Concern about Supplement | 2 | 0
Not completed — Inconvenience | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Began hypertension medication | 1 | 0
Not completed — Began cancer treatments | 1 | 0
Not completed — Moved from area | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pine Bark Extract: 200 mg Flavangenol delivered once per day orally. Flavangenol is a brand of Pine Bark Extract manufactured by Toyo Shinyaku of Saga, Japan. Dosage delivered as four tablets 50 mg each; 4 tablets taken in the morning daily. Pine Bark Extract (Flavangenol�) : Flavangenol 200 mg per day. Dosage delivered as four tablets, 50 mg per tablet, taken once per day orally for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Pine Bark Extract | Placebo | Total
Number analyzed (Participants) | 64 | 66 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 55 | 106
  >=65 years | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (9.8) | 53.9 (12.0) | 55.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 39 | 43 | 82

OUTCOME MEASURES:

1. Primary Outcome: Combined Change in Systolic and Diastolic Blood Pressures From Baseline to Week 12.
Description: Mean at Week 12 observation minus mean at Baseline observation.
Time Frame: three months
Population: The data was analyzed on an intent-to-treat basis, with the last observation collected carried forward for participants with missing data at follow-up.
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Pine Bark Extract | Placebo
Number analyzed (Participants) | 64 | 66
mm Hg | -1.0 [-4.2 to 2.1] | -1.9 [-5.5 to 1.7]

2. Secondary Outcome: Total Cholesterol
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Pine Bark Extract (Net Change): 200 mg Flavangenol delivered once per day orally. Flavangenol is a brand of Pine Bark Extract manufactured by Toyo Shinyaku of Saga, Japan. Dosage delivered as four tablets 50 mg each; 4 tablets taken in the morning daily.
  Pine Bark Extract (Flavangenol®) : Flavangenol 200 mg per day. Flavangenol is a brand of pine bark extract manufactured by Toyo Shinyaku of Saga, Japan.
  Dosage delivered as four tablets, 50 mg per tablet, taken once per day orally for 12 weeks.
- Placebo (Net Change): Placebo delivered as four tablets matching the active product; four tablets taken daily orally.
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 60 | 62
mg/dL | 5.4 (17.5) | -2.0 (23.7)
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = 7.3, 95% CI 2-sided [-0.1 to 14.9]

3. Secondary Outcome: LDL
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 60 | 62
mg/dL | 3.3 (16.6) | -1.1 (19.7)
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = 4.4, 95% CI 2-sided [-2.1 to 10.8]

4. Secondary Outcome: HDL
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 60 | 62
mg/dL | -0.9 (6.0) | -1.3 (5.6)
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = 0.4, 95% CI 2-sided [-1.7 to 2.5]

5. Secondary Outcome: Triglycerides
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up).
Time Frame: three months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 60 | 62
mg/dL | 17.2 (50.6) [-0.1 to 0.3] | -1.0 (63.0) [-0.0 to 0.1]
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = 18.2, 95% CI 2-sided [-2.3 to 38.7]

6. Secondary Outcome: LDL Particle Size
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 59 | 62
nm | 31.4 (200.2) | 28.5 (248.5)
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.1 to 0.3]

7. Secondary Outcome: HDL Particle Size
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 59 | 62
nm | 1.0 (3.1) | 0.0 (4.2)
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.0 to 0.1]

8. Secondary Outcome: Lipoprotein A
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up). Calculated as (Pinebark_Followup - Pinebark_Baseline) - (Placebo_Follow-up - Placebo_Baseline)
Time Frame: three months
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 59 | 60
nmol/L | -1.3 (10.3) [-6.8 to 0.5] | 1.8 (10.0)
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = -3.2, 95% CI 2-sided [-6.8 to 0.5]

9. Secondary Outcome: C-reactive Protein
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up).
Time Frame: three months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 60 | 63
nmol/L | -0.2 (2.56) [-1.5 to 0.5] | 0.3 (2.9)
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.5 to 0.5]

10. Secondary Outcome: Body Mass Index
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up).
Time Frame: three months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 60 | 62
kg/m^2 | 0.1 (0.4) [0.0 to 0.4] | -0.1 (0.6)
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = 0.2, 95% CI 2-sided [0.0 to 0.4]

11. Secondary Outcome: Weight
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: lb
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 60 | 62
lb | 0.6 (3.1) | -0.6 (3.4)
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = 1.2, 95% CI 2-sided [0.1 to 2.4]

12. Secondary Outcome: Fasting Blood Glucose
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up).
Time Frame: three months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 59 | 62
mg/dL | -1.0 (9.8) [-4.4 to 2.3] | 0.1 (8.7)
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = -1.0, 95% CI 2-sided [-4.4 to 2.3]

13. Secondary Outcome: Fasting Insulin
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up).
Time Frame: three months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 60 | 62
mg/dL | 0.2 (4.2) [-0.9 to 2.5] | -0.6 (5.2)
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = 0.8, 95% CI 2-sided [-0.9 to 2.5]

14. Secondary Outcome: Hemoglobin A1c
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up).
Time Frame: three months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 58 | 62
mg/dL | -0.0 (0.2) [-0.1 to 0.1] | -0.0 (0.2)
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.1 to 0.1]

15. Secondary Outcome: ALT/SGPT
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up).
Time Frame: three months
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 60 | 62
u/L | 0.8 (15.11) [-1.6 to 9.3] | -3.0 (15.28)
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = 3.8, 95% CI 2-sided [-1.6 to 9.3]

16. Secondary Outcome: AST/SGOT
Description: Net change in secondary outcomes from Baseline to 12 Weeks (Follow-up).
Time Frame: three months
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Pine Bark Extract (Net Change) | Placebo (Net Change)
Number analyzed (Participants) | 60 | 62
u/L | 0.2 (4.9) [-3.4 to 0.8] | 1.4 (6.8)
Statistical Analysis 1: Comparison: Pine Bark Extract (Net Change) vs Placebo (Net Change); Test type: Superiority or Other; Mean Difference (Net) = -1.3, 95% CI 2-sided [-3.4 to 0.8]

ADVERSE EVENTS:
Arm/Group | Pine Bark Extract | Placebo
Serious Adverse Events (participants affected / at risk) | 1/64 | 2/66
Other Adverse Events (participants affected / at risk) | 24/64 | 29/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pine Bark Extract (N=64) | Placebo (N=66)
Hospitalized (Surgical and medical procedures) | 1 (1) | 0 (0) — Hip Surgery
Emergency Department (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — Dislocated toe; Received tetanus booster after stepping on a nail
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pine Bark Extract (N=64) | Placebo (N=66)
Gastrointestinal Discomfort (week 3) (Gastrointestinal disorders) | 12 (12) | 9 (9)
Gastrointestinal Discomfort (week 6) (Gastrointestinal disorders) | 8 (8) | 3 (3)
Nause (week 12) (Gastrointestinal disorders) | 6 (6) | 1 (1)
Dizziness (week 3) (Nervous system disorders) | 1 (1) | 5 (5)
Dizziness (week 12) (Nervous system disorders) | 3 (3) | 7 (7)
Headache (week 12) (Nervous system disorders) | 8 (8) | 13 (13)
Sleepiness (week 12) (General disorders) | 5 (5) | 12 (12)
Insomnia (week 6) (Nervous system disorders) | 4 (4) | 11 (11)
Increased Perspiration (week 6) (General disorders) | 5 (5) | 1 (1)
Other (week 6) (General disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No